CLINICAL TRIAL: NCT04461600
Title: A Phase 2, Multi-center, Open-label, Single Arm Study of AL101 Monotherapy in Patients With Notch Activated Triple Negative Breast Cancer
Brief Title: A Study of AL101 Monotherapy in Patients With Notch Activated Triple Negative Breast Cancer
Acronym: TENACITY
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Ayala Pharmaceuticals, Inc, (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL-TNBC-01
Record Dates: First submitted 2020-06-29; First posted 2020-07-08 (Actual); Results first posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-01

CONDITIONS: Triple Negative Breast Cancer
Keywords: TNBC, Notch activated
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AL101 (Experimental): The study included a lead-in cohort with 6 subjects at 6mg AL101 weekly. 13 additional patients were treated with 4mg AL101 weekly.
  Interventions: Drug: AL101

INTERVENTIONS:
Drug: AL101 — AL101 is an inhibitor of gamma secretase-mediated Notch signaling.

SUMMARY:
The current study is designed to evaluate the efficacy and safety of AL101 monotherapy in subjects with Notch-activated recurrent or metastatic TNBC; Notch activation will be determined by a Next Generation Sequencing (NGS) test.

ELIGIBILITY:
Inclusion Criteria:

1. Male of female subjects who are at least 18 years of age (inclusive) at the time of signing the Informed Consent Form (ICF).
2. Have at least one measurable lesion per RECIST v1.1.
3. Have formalin-fixed paraffin-embedded (FFPE) tissue available from a metastatic lesion; a tumor block or 25 unstained slides from an archived (within 2 years) or fresh tumor samples (core or punch needle biopsy) are acceptable.
4. Documented tumor progression following no more than 3 lines of systemic chemotherapy, PARP inhibitor therapy or immunotherapy for metastatic disease, as appropriate. Of note, neoadjuvant and adjuvant therapy will not count as prior lines of therapy.
5. Histologically confirmed diagnosis of inoperable locally advanced or metastatic TNBC defined as ER and progesterone receptor staining <10%, and HER2 negative defined as IHC 0 to 1+
6. Documented Notch activation from tumor biopsy results from within the last 2 years from a commercially available NGS assay, LDT or other validated IUO clinical trial assay.
7. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test.

Exclusion Criteria:

1. A known additional malignancy that is progressing or requires active treatment that is considered medically active and may interfere in the ability to detect responses in this subject. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that have undergone potentially curative therapy or in situ cervical cancer.
2. BC that, in the opinion of the investigator, is considered amenable to potentially curative treatment.
3. Symptomatic central nervous system (CNS) metastases.
4. Current or recent (within 2 months of IP administration) gastrointestinal (GI) disease or disorders that increase the risk of diarrhea, such as inflammatory bowel disease and Crohn's disease.
5. Developed immune-mediated colitis with immunotherapy unless resolved to G1 or lower and without requirement of steroid treatment for at least 14 days prior to first dose of IP.
6. Peripheral neuropathy Grade 2 for at least 14 days prior to first dose of IP.
7. Evidence of uncontrolled, active infection, requiring systemic anti-bacterial, anti-viral or anti-fungal therapy ≤7 days prior to administration of IP such as known active infection with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
8. Unstable or severe uncontrolled medical condition (e.g., unstable cardiac or pulmonary function or uncontrolled diabetes) or any important medical illness or abnormal laboratory finding that would, in the investigator's judgment, increase the risk to the subject associated with his or her participation in the study.
9. Eastern Cooperative Oncology Group (ECOG) performance status ≥2.
10. Abnormal organ and marrow function defined as:

    1. neutrophils <1000/mm3,
    2. platelet count <75,000/mm3,
    3. hemoglobin <8 g/dL,
    4. total bilirubin >1.5 upper limit of normal (ULN) (except known Gilbert's syndrome whereby the total bilirubin must be < 5 mg/dL),
    5. aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >2.5 ULN OR >5 ULN for subjects with liver metastases,
    6. creatinine clearance (CrCl) <50 mL/min (calculation of CrCl will be based on acceptable institution standard),
    7. uncontrolled triglyceride ≥Grade 2 elevations per CTCAE v5.0 (>300 mg/dL or >3.42 mmol/L).
11. Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
12. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥480 msec.
13. Completed palliative radiation therapy < 7 days prior to initiating IP.
14. Prior treatment with gamma secretase inhibitors.
15. Last chemotherapy, biologic, or investigational therapy agent at least 4 weeks or 5 half-lives (whichever is shorter) prior to initiating IP; at least 6 weeks if the last regimen included BCNU or mitomycin C. Prior treatment with investigational monoclonal antibody will be reviewed case-by-case by the Sponsor.
16. Receiving chronic systemic steroid therapy (in dosing exceeding 10 mg/day of prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of IP. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.
17. Use of strong inhibitors of CYP3A4 within 1 week or 5 half-lives (whichever is longer) or strong inducers of CYP3A4 within 2 weeks or 5 half-lives (whichever is longer).
18. Life expectancy is less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andres Gutierrez, MD, PhD, Study Director — Executive Vice President & Chief Medical Officer
Locations (29):
- United States (17):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - University of California at San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Comprehensive Hematology Oncology, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - The University of Chicago, Chicago, Illinois
  - Carle Clinic, Urbana, Illinois
  - University of Louisville- James Brown Cancer Center, Louisville, Kentucky
  - Maryland Oncology Hematology, Columbia, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Central Cancer Care, Bolivar, Missouri
  - Memorial Sloan Kettering Cancer Center (MSKCC), New York, New York
  - University Health Cleveland Medical Center, Cleveland, Ohio
  - Charleston Oncology, Charleston, South Carolina
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - UZ Leuven, Leuven
- Israel (5):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Hospital, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
- Spain (3):
  - Vall d'Hebron University Hospital, Barcelona
  - Institut Català d'Oncologia, Barcelona
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
- United Kingdom (2):
  - The Christie Hospital, Manchester, England
  - University Hospital of Edinburgh, Edinburgh, Scotland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AL101 4mg: AL101 is an inhibitor of gamma secretase-mediated Notch signaling. 4mg of AL101 was administered using an IV infusion pump over 60 minutes, once a week.
- AL101 6mg: AL101 is an inhibitor of gamma secretase-mediated Notch signaling. 6mg of AL101 was administered using an IV infusion pump over 60 minutes, once a week.
Period: Overall Study
Arm/Group | AL101 4mg | AL101 6mg
Started | 12 | 6
Completed | 6 | 0
Not Completed | 6 | 6
Not completed — Death | 6 | 5
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AL101 4mg | AL101 6mg | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 6 | 17
  >=65 years | 1 | 0 | 1
Age, Continuous [Median (Full Range); unit: years] | 48 [30 to 87] | 45 [36 to 55] | 48 [30 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 19 patients were enrolled, only 18 were treated.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 1 | 1
    White | 9 | 5 | 14
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Belgium | 1 | 0 | 1
  United States | 5 | 5 | 10
  Israel | 1 | 1 | 2
  Spain | 5 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as partial response (PR) + complete response (CR) as assessed by the investigator based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 for target lesions assessed by MRI.
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 12 month
Population: Efficacy Evaluable Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | AL101 6mg | AL101 4mg
Number analyzed (Participants) | 3 | 10
Participants | 0 | 0

2. Secondary Outcome: Clinical Benefit Response Rate (CBR)
Description: Clinical benefit response rate (CBR) is defined as complete response (CR) + partial response (PR) + stable disease (SD) by investigator review based on RECIST v1.1 for target lesions assessed by MRI.
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Stable Disease (SD): Neither sufficient shrinkage (at least 30%) to qualify for PR nor sufficient increase (more than 20%) to qualify for PD, taking as reference the smallest sum diameters.
Time Frame: 12 month
Population: Efficacy Evaluable Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | AL101 6mg | AL101 4mg
Number analyzed (Participants) | 3 | 10
Participants | 1 | 3

3. Secondary Outcome: Duration of Response (DOR) by Investigator Review Based on RECIST v1.1
Description: Duration of response (DOR) is defined as the time from randomization to disease progression or death in patients who achieve complete or partial response.
Time Frame: 12 month
Population: Duration of response data was not collected as there were no patients with either CR or PR
Arm/Group | AL101 6mg | AL101 4mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year and 3 months
Description: The analysis was done on the safety population which consists of 18 patients (6 patients in the 6mg arm, and 12 patients in the 4mg arm)
Groups:
- AL101 6mg: AL101 is an inhibitor of gamma secretase-mediated Notch signaling.
  .
- AL101 4mg: AL101 is an inhibitor of gamma secretase-mediated Notch signaling.
Arm/Group | AL101 6mg | AL101 4mg
All-Cause Mortality (participants affected / at risk) | 5/6 | 6/12
Serious Adverse Events (participants affected / at risk) | 5/6 | 2/12
Other Adverse Events (participants affected / at risk) | 6/6 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AL101 6mg (N=6) | AL101 4mg (N=12)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AL101 6mg (N=6) | AL101 4mg (N=12)
Diarrhoea (Gastrointestinal disorders) | 5 | 5
Nausea (Gastrointestinal disorders) | 3 | 5
Vomiting (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 2 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1
Eructation (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 2 | 5
Asthenia (General disorders) | 0 | 4
Pyrexia (General disorders) | 1 | 3
Influenza like illness (General disorders) | 0 | 2
Mucosal inflammation (General disorders) | 0 | 2
Pain (General disorders) | 0 | 2
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Device related thrombosis (General disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Localised oedema (General disorders) | 0 | 1
Mucosal dryness (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 6
Dizziness (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 0 | 2
Anosmia (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Dystonia (Nervous system disorders) | 0 | 1
Taste disorder (Nervous system disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatine increased (Investigations) | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 3
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Cystitis (Infections and infestations) | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 2
Acute sinusitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Sputum purulent (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Cushing's syndrome (Endocrine disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT04461600/Prot_SAP_000.pdf